CLINICAL TRIAL: NCT05141773
Title: Computer-assisted Adenoma Detection Coloscopy With Endo-AID Artificial Intelligence System and Endocuff Versus Endocuff Assisted Colonoscopy: a Randomized Controlled Trial
Brief Title: Artificial Intelligence Aid Systems and Endocuff in Colorectal Adenoma Detection
Acronym: CUFFAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Computer aid colonoscopy
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Adenoma Detection Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Computed adenoma detection system (CADe) and Endocuff (Experimental): CADe system can detect in the screen suspicion areas of adenomatous polyps. This is an additional help for the endoscopist for the detection of lesions. Endocuff increases the colonic surface examinated
  Interventions: Device: Computed adenoma detection system (CADe) plus endocuff
- Control group (Endocuff) (Active Comparator): Endocuff increases the colonic surface examinated
  Interventions: Device: Endocuff

INTERVENTIONS:
Device: Computed adenoma detection system (CADe) plus endocuff — This is a computed system that helps the endoscopist to increase the detection of colorectal polyps. An add-on device (Endocuff) is also incorporated to the tip of the colonoscope
  Arms: Computed adenoma detection system (CADe) and Endocuff
Device: Endocuff — An add-on device (Endocuff) is also incorporated to the tip of the colonoscope
  Arms: Control group (Endocuff)

SUMMARY:
The main purpose of the study to evaluate the usefulness of the Endo-AID artificial intelligence system combined with endocuff compared with endocuff in the detection of colorectal adenomas in consecutive patients for outpatient colonoscopy.

The secondary aims were:

* To evaluate the benefit of Endo-AID and endocuff in adenoma detection rate by comparing endoscopists with high and low adenoma detection rate.
* To evaluate serrated detection rate, advanced adenoma detection rate, adenoma detection rate according to the size (<= 5mm, 6-9mm,> = 10mm) and number of adenomas by colonoscopy. Stratification by location and morphology.

DETAILED DESCRIPTION:
Guidelines have been established regarding artificial intelligence (AI) applied to gastrointestinal endoscopy. Regarding the priority uses for their development, there are applications that improve vision, placing computer-assisted lesion detection (CADe) as one of the most necessary priorities, given the importance of colorectal cancer screening (CRC) and post-polypectomy surveillance. The evaluation of these systems in different clinical practices and patient groups has been recommend. In this regard, studies in the western population are limited and have been carried out by expert endoscopists. It has not been evaluated comparing with other strategies such as add-on devices. In addition, there are no studies with the recent CADe Endo-AID system (Olympus Corp. Tokyo).

The main purpose of the study is to evaluate the usefulness of the Endo-AID artificial intelligence system with endocuff in the detection of colorectal adenomas in consecutive patients for outpatient colonoscopy compared with standard colonoscopy with endocuff. In addition, the benefit of the CADe system will be assessed according to the endoscopist ADR.

A randomized controlled trial will be carried out in consecutive outpatients meeting the inclusion criteria and none of the exclusion criteria. Patients with be randomized to one of the two groups: CADe system with endocuff and standard colonoscopy with endocuff.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients referred for outpatient colonoscopy

Exclusion Criteria:

* Colonic resection
* Taking anticoagulants or antiaggregants that contraindicate the performance of therapy
* Patients with a recent colonoscopy (<6 months) of good quality (e.g. cited for endoscopic therapy)
* IBD
* Patients with incomplete colonoscopy
* Patients with inadequate preparation using the Boston Colonic Preparation Scale (BBPS). A cleaning quality of less than 2 points in any of the 3 colonic sections will be considered inadequate.
* Patients with polyposis syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 1 year
  (number of colonoscopies with adenoma/number of colonoscopies)

SECONDARY OUTCOMES:
Serrated detection rate | 1 year
  (number of colonoscopies with serrated adenoma/number of colonoscopies)
Advanced adenoma detection rate | 1 year
  (number of colonoscopies with advanced adenomas/number of colonoscopies)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Z García, MD, PhD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, SANTA CRUZ DE TENERIFE, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngu WS, Bevan R, Tsiamoulos ZP, Bassett P, Hoare Z, Rutter MD, Clifford G, Totton N, Lee TJ, Ramadas A, Silcock JG, Painter J, Neilson LJ, Saunders BP, Rees CJ. Improved adenoma detection with Endocuff Vision: the ADENOMA randomised controlled trial. Gut. 2019 Feb;68(2):280-288. doi: 10.1136/gutjnl-2017-314889. Epub 2018 Jan 23. PMID 29363535
- [Background] Repici A, Badalamenti M, Maselli R, Correale L, Radaelli F, Rondonotti E, Ferrara E, Spadaccini M, Alkandari A, Fugazza A, Anderloni A, Galtieri PA, Pellegatta G, Carrara S, Di Leo M, Craviotto V, Lamonaca L, Lorenzetti R, Andrealli A, Antonelli G, Wallace M, Sharma P, Rosch T, Hassan C. Efficacy of Real-Time Computer-Aided Detection of Colorectal Neoplasia in a Randomized Trial. Gastroenterology. 2020 Aug;159(2):512-520.e7. doi: 10.1053/j.gastro.2020.04.062. Epub 2020 May 1. PMID 32371116
- [Background] Aziz M, Haghbin H, Gangwani MK, Sharma S, Nawras Y, Khan Z, Chandan S, Mohan BP, Lee-Smith W, Nawras A. Efficacy of Endocuff Vision compared to first-generation Endocuff in adenoma detection rate and polyp detection rate in high-definition colonoscopy: a systematic review and network meta-analysis. Endosc Int Open. 2021 Jan;9(1):E41-E50. doi: 10.1055/a-1293-7327. Epub 2021 Jan 1. PMID 33403235
- [Background] Ashat M, Klair JS, Singh D, Murali AR, Krishnamoorthi R. Impact of real-time use of artificial intelligence in improving adenoma detection during colonoscopy: A systematic review and meta-analysis. Endosc Int Open. 2021 Apr;9(4):E513-E521. doi: 10.1055/a-1341-0457. Epub 2021 Mar 17. PMID 33816771
- [Background] Barua I, Vinsard DG, Jodal HC, Loberg M, Kalager M, Holme O, Misawa M, Bretthauer M, Mori Y. Artificial intelligence for polyp detection during colonoscopy: a systematic review and meta-analysis. Endoscopy. 2021 Mar;53(3):277-284. doi: 10.1055/a-1201-7165. Epub 2020 Sep 29. PMID 32557490
- [Background] Hassan C, Spadaccini M, Iannone A, Maselli R, Jovani M, Chandrasekar VT, Antonelli G, Yu H, Areia M, Dinis-Ribeiro M, Bhandari P, Sharma P, Rex DK, Rosch T, Wallace M, Repici A. Performance of artificial intelligence in colonoscopy for adenoma and polyp detection: a systematic review and meta-analysis. Gastrointest Endosc. 2021 Jan;93(1):77-85.e6. doi: 10.1016/j.gie.2020.06.059. Epub 2020 Jun 26. PMID 32598963